CLINICAL TRIAL: NCT03159156
Title: Respiration and Applied Tension Strategies to Reduce Vasovagal Reactions to Blood Donation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: MOP-133459
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Syncope, Vasovagal
MeSH Terms: conditions — Syncope, Vasovagal | interventions — arcA protein, E coli

STUDY DESIGN:
Intervention Model Description: The primary goal is to examine the role of hyperventilation in blood donation-related vasovagal reactions and whether breathing is influenced by two treatments (alone and in combination) for reactions. The study will examine the clinical impact of these treatments but this is not the primary goal of the project.
Masking Description: Behavioral procedures that cannot be masked to participant or others.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blood Donation As Usual (No Intervention): Volunteer blood donors complete assessment materials, including assessment of respiratory activity, but otherwise undergo the typical blood donation procedure.
- Applied Tension (Experimental): Participants are taught a simple muscle tensing technique with a brief video presented on a notebook computer before giving blood. They are asked to engage in repeated gentle 5-sec on, 5-sec off cycles of whole body isometric muscle tension before and while giving blood.
  Interventions: Behavioral: Applied Tension
- Respiration Control (Experimental): Participants are taught a simple respiration control technique with a brief video presented on a notebook computer before giving blood. They are asked to breathe in a gentle shallow but regular fashion aimed at reducing risk for hyperventilation before and while giving blood.
  Interventions: Behavioral: Respiration Control
- Applied Tension/Respiration Control (Experimental): Participants are asked to practice both Applied Tension and Respiration Control before and while giving blood.
  Interventions: Behavioral: Applied Tension/Respiration Control

INTERVENTIONS:
Behavioral: Applied Tension — Described above.
  Arms: Applied Tension
Behavioral: Respiration Control — Described above.
  Arms: Respiration Control
Behavioral: Applied Tension/Respiration Control — Described above.
  Arms: Applied Tension/Respiration Control

SUMMARY:
For a number of years, researchers have examined the effects of the muscle-tensing technique, Applied Tension (AT), on blood donation-related vasovagal symptoms and donor retention. AT was developed originally to reduce symptoms and avoidance behaviour in people with strong fears of blood and needles (phobics). It was based on the idea that exercise-related increases in blood pressure might be able to counteract the effects of stimuli that lead to a decrease in delivery of blood to the brain. AT was adapted for non-phobic blood donors and significant reductions in self-reported vasovagal symptoms and the need for nurse-initiated treatment as well as increases in donor retention were observed in some groups.

That said, individual response to AT is quite variable. This is probably related to recent research indicating that exercise-related maintenance of heart rate and blood pressure plays only a minor role in reducing vasovagal symptoms. Rather, AT appears to be working at least in part by regulating breathing and reducing the possibility of hyperventilation. Pilot results suggest that a novel intervention aimed specifically at breathing may be more effective and reliable than traditional AT. To evaluate this idea, 408 blood donors at mobile clinics in colleges and universities will be assigned randomly to four conditions. In brief, 5-minute preparation sessions using a notebook computer, donors will either learn a respiration control technique to avoid hyperventilation, AT, both, or neither. As a manipulation check and also a means of examining mechanisms of the interventions, e.g., the possibility that AT may work by regulating breathing and CO2, participants will wear non-invasive portable capnometers while they are giving blood. Outcome will also be assessed by self-report of vasovagal symptoms, observational data, and number of return visits to a blood clinic in the following year verified by the provincial blood collection agency, Héma-Québec. As a secondary aim, the research will examine possible moderating effects of pre-donation anxiety and sex.

The development of simple, effective approaches to reduce vasovagal symptoms during blood donation has the potential to improve the blood donation experience and blood donor retention as well as encourage people who have never given blood to consider the procedure. It will also improve medical and dental care more generally given the use of needles in so many procedures.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer blood donors.

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 408 (Estimated)
Dates: Start 2015-09-15 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in End Tidal CO2 | change in mean value during the pre-donation waiting period (registration to going to chair, approximately 30 minutes) to the mean value in the donation chair (approximately 15 minutes)
  assessed by ambulatory monitor (capnometer)
Change in Respiration Rate | change in mean value during the pre-donation waiting period (registration to going to chair, approximately 30 minutes) to the mean value in the donation chair (approximately 15 minutes)
  assessed by ambulatory monitor (capnometer)
Blood Donation Reactions Inventory | completed in the recovery area, approximately 15 minutes after blood donation
  questionnaire assessing presyncopal vasovagal symptoms
Research Assistant Observations | during blood donation
  participant anxiety, fainting, whether or not treatment for a vasovagal response required, etc., noted by a research assistant

SECONDARY OUTCOMES:
Change in Spielberger State Anxiety Scale Score | completed just after registering at the clinic and also in the recovery area, approximately 15 minutes after blood donation, to assess change in anxiety
  self-report questionnaire
Medical Fears Survey | completed in the recovery area, approximately 15 minutes after blood donation
  self-report questionnaire
Change in Systolic Blood Pressure | measured just after registering at the clinic and also in the recovery area, approximately 15 minutes after blood donation, to assess change in blood pressure
  in mmHg
Change in Diastolic Blood Pressure | measured just after registering at the clinic and also in the recovery area, approximately 15 minutes after blood donation, to assess change in blood pressure
  in mmHg
Change in Heart Rate | measured just after registering at the clinic and also in the recovery area, approximately 15 minutes after blood donation, to assess change in heart rate
  in bpm
Blood Donor Return | one year after participating in the study
  number of times the donor returns to give blood again in a one-year time frame as reported by Hema-Quebec

CONTACTS AND LOCATIONS:
Overall Officials: Blaine Ditto, PhD, Principal Investigator — Professor
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided